CLINICAL TRIAL: NCT07008274
Title: Laparoscopic Sleeve Gastrectomy-Induced Decline in Plasma Asprosin and Its Association With Metabolic Recovery
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Director, Northern Jiangsu People's Hospital
Other Study IDs: NorthernJiangsu123
Record Dates: First submitted 2025-05-11; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Morbid
Keywords: bariatric surgery; asprosin
MeSH Terms: conditions — Obesity, Morbid; Arachnodactyly | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- surgery: surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — laparoscopic sleeve gastrectomy

SUMMARY:
the present study aimed to systematically assess the changes in plasma asprosin levels at 3, 6, and 12 months after LSG, to explore the relationships between asprosin dynamics and key metabolic parameters, including body mass index (BMI), fasting glucose, insulin resistance assessed by the homeostasis model (HOMA-IR), and lipid profiles, and to compare asprosin concentrations between bariatric patients and healthy normal-weight controls.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years;
2. body mass index (BMI) ≥37.5 kg/m², or BMI ≥32.5 kg/m² with at least one obesity-related comorbidity;
3. availability of complete clinical data and stored plasma samples at preoperative baseline and at 3, 6, and 12 months postoperatively.

Exclusion Criteria:

1. history of prior bariatric or gastrointestinal surgery;
2. active malignancy, chronic inflammatory or infectious disease, or severe hepatic or renal dysfunction;
3. pregnancy during the study period;
4. incomplete clinical or biochemical data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults with obesity (BMI ≥37.5 kg/m², or ≥32.5 kg/m² with metabolic comorbidities such as type 2 diabetes, hypertension, or dyslipidemia), aged 18-65 years, undergoing laparoscopic sleeve gastrectomy at a single tertiary hospital in China. Healthy normal-weight controls (BMI 18.5-23.9 kg/m²) without metabolic disorders were also recruited for baseline comparison.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma asprosin levels at 3, 6, and 12 months | 1 year

SECONDARY OUTCOMES:
BMI at 3, 6, and 12 months | 1 year

OTHER OUTCOMES:
Insulin resistance (HOMA-IR) at 3, 6, and 12 months | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shuai Zhao, Yangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: No